CLINICAL TRIAL: NCT05461742
Title: Pilot Testing an Innovative Physical Activity Intervention for Parents
Brief Title: Pilot Testing an Innovative Physical Activity Intervention for Parents Attending Their Children's Sport Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022003323; U54GM115677 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Physical Inactivity
Keywords: physical activity; exercise; disparities; parents; mothers
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention (Experimental): All participants will receive a physical activity intervention consisting of goal setting, in-person physical activity sessions, and written materials.
  Interventions: Behavioral: Physical activity intervention

INTERVENTIONS:
Behavioral: Physical activity intervention — While the final content and structure of the intervention will be informed by community advisory board, participants will receive a culturally adapted, Social Cognitive Theory and Transtheoretical Model-based PA intervention. The evidence-based, theory guided aerobic physical activity intervention will systematically build upon the investigators' prior studies and includes the following components: goal setting, in-person physical activity sessions, and written materials.

SUMMARY:
The intervention aims to increase physical activity, an important health behavior, in a high-risk sample (i.e., Black and Hispanic/Latino mothers). The study builds on the investigators' previous work by adapting an evidence-based theory guided physical activity intervention to be implemented in a community setting mothers regularly spend time for their children's extracurricular activities, circumventing barriers commonly cited by racial/ethnic minority mothers (e.g., other responsibilities, time barriers, transportation, and childcare). The investigators will partner with a local youth sports organization to adapt and deliver a physical activity intervention to mothers during practice. They aim to convene a community advisory board of coaches and parents to enhance participant acceptability and work through any feasibility issues with implementation. The investigators will then conduct an open pilot trial of the physical activity intervention administered to mothers during their children's sports practices. They will assess feasibility, acceptability, and examine the effects of the intervention on mothers' physical activity. The investigators hypothesize that mothers in the intervention will increase their physical activity.

DETAILED DESCRIPTION:
The intervention aims to increase physical activity, an important health behavior, in a high-risk sample (i.e., Black and Hispanic/Latino mothers). As physical activity impacts risk for obesity and related chronic diseases (Type II diabetes, heart disease, etc.), national guidelines recommend that adults engage in 150 minutes of moderate intensity aerobic activity per week. More than half of adults in Rhode Island do not meet this recommendation, and racial and ethnic minorities are disproportionately burdened by obesity, and often exhibit suboptimal physical activity-related behaviors. Racial/ethnic minority mothers may be at particularly high risk for obesity, not just because of weight gain in the perinatal period, but because the transition to parenthood, often accompanied by sleep disruption and decreased physical activity, is a critical window for adult health and can shape health trajectories in midlife. Further, mothers often report too many responsibilities and prioritizing their children's needs as barriers to engaging in more physical activity. Racial/ethnic minority mothers are especially likely to report lack of time as a barrier to being more physically active. Interventions are therefore needed that address specific barriers among this high-risk population. The study builds on the investigators' previous work by adapting an evidence-based theory guided physical activity intervention to be implemented in a community setting mothers regularly spend time for their children's extracurricular activities, circumventing barriers commonly cited by racial/ethnic minority mothers (e.g., other responsibilities, time barriers, transportation, and childcare). They will partner with a local youth sports organization to adapt and deliver a physical activity intervention to mothers during practice.

The investigators aim to convene a community advisory board of coaches and parents to enhance participant acceptability and work through any feasibility issues with implementation. The community advisory board will include coaches and mothers from our partner organization, the local youth football and cheerleading organization. The investigators will engage the community advisory board to partner with us in adapting and refining the intervention. Prior to the intervention, the community advisory board will inform the structure of the in-person physical activity sessions. They will continue to meet with the community advisory board over the study period to gain feedback around implementation and inform changes for a subsequent grant a fully powered randomized controlled trial.

The second aim is to conduct an open pilot trial of the physical activity intervention administered to mothers during their children's sports practices. The investigators aim to recruit 45 mothers to participate in a single arm pre-test, post-test design pilot study of the intervention, which will last for 8 weeks. They plan to demonstrate feasibility of recruitment, retention, and data collection procedures, and acceptability of the intervention using specified benchmarks. All participants will complete exit surveys at the end of the intervention, with 15 participants invited to also complete an in depth interview. The investigators will also examine within-person changes in minutes of moderate to vigorous physical activity over time (e.g., from baseline to intervention end (8-weeks), and at 1-month follow up), as well as intervention dose effects (e.g., number of physical activity sessions attended/week) on change in minutes of moderate to vigorous physical activity.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Identifying as female
* Having (or being the primary caregiver of) a child who is a current member of one of the partner organization's teams/squads
* Having email access
* Being able to speak and read English or Spanish.

Exclusion Criteria:

* For safety reasons, participants who do not pass the Physical Activity Readiness Questionnaire, a community screener used to detect those who may be at risk when increasing their physical activity, will be excluded from participating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as female
Enrollment: 35 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tayla von Ash, ScD, MPH, Principal Investigator — Brown University School of Public Health
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity Intervention
Started | 35
Completed | 33
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Physical Activity Intervention
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.18 (5.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 2
  More than one race | 8
  Unknown or Not Reported | 16

OUTCOME MEASURES:

1. Primary Outcome: Moderate to Vigorous Physical Activity (Minutes/Week)
Description: Assessed using the 7-Day Physical Activity Recall Interview
Time Frame: Change from baseline to end of treatment (8 weeks)
Population: Due to missing data, the number of participants analyzed is smaller than recruited.
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Physical Activity Intervention
Number analyzed (Participants) | 20
minutes/week | 26.10 (155.28)

ADVERSE EVENTS:
Time Frame: 2 months
Description: All-Cause Mortality, Serious, or Other (non-serious) Adverse Events were monitored/assessed
Arm/Group | Physical Activity Intervention
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/42/NCT05461742/Prot_SAP_000.pdf